CLINICAL TRIAL: NCT03449511
Title: Aromatherapy: An Integrative Option for Symptom Management in Cancer Care
Brief Title: Aromatherapy for Integrated Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Julie Ryan Wolf, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 71162
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ginger aromatherapy (Active Comparator): Ginger essential oil (GIN-106) in an aromatherapy inhaler. Subject will take 3 sniffs of the inhaler four times daily (morning, noon, evening, bedtime) for 7 consecutive days during two chemotherapy cycles.
  Interventions: Other: Ginger aromatherapy
- Orange aromatherpy (Active Comparator): Orange essential oil (ORG-114) in an aromatherapy inhaler. Subject will take 3 sniffs of the inhaler four times daily (morning, noon, evening, bedtime) for 7 consecutive days during two chemotherapy cycles.
  Interventions: Other: Orange aromatherapy
- Lavender aromatherapy (Active Comparator): Lavender essential oil (LAV-110) in an aromatherapy inhaler. Subject will take 3 sniffs of the inhaler four times daily (morning, noon, evening, bedtime) for 7 consecutive days during two chemotherapy cycles.
  Interventions: Other: Lavender aromatherapy
- Jojoba aromatherapy (Placebo Comparator): Jojoba oil in an aromatherapy inhaler. Subject will take 3 sniffs of the inhaler four times daily (morning, noon, evening, bedtime) for 7 consecutive days during two chemotherapy cycles. One drop of jojoba oil is on the other three aromatherapy inhalers. Jojoba oil is a "carreir oil" for essential oils which will be used as a comparator and placebo in this study.
  Interventions: Other: Jojoba aromatherapy

INTERVENTIONS:
Other: Ginger aromatherapy — Three sniffs of aromatherapy inhaler four times daily for seven days.
  Arms: Ginger aromatherapy
Other: Orange aromatherapy — Three sniffs of aromatherapy inhaler four times daily for seven days.
  Arms: Orange aromatherpy
Other: Lavender aromatherapy — Three sniffs of aromatherapy inhaler four times daily for seven days.
  Arms: Lavender aromatherapy
Other: Jojoba aromatherapy — Three sniffs of aromatherapy inhaler four times daily for seven days.
  Arms: Jojoba aromatherapy

SUMMARY:
The purpose of this clinical trial is to determine the feasibility and effectiveness of aromatherapy in relief of commonly reported symptoms in cancer patients undergoing chemotherapy. Aromatherapy is a noninvasive, minimal risk intervention that could potentially alleviate the severity of treatment-related symptoms. This study will evaluate the ability of four aromatherapy scents (ginger, lavender, orange, jojoba) to reduce the severity of seven chemotherapy-induced symptoms (nausea, vomiting, pain, anxiety/distress, fatigue, sleep difficulties, and lack of appetite). Jojoba oil is a " carrier oil" and will act as a placebo comparator in this study. Jojoba oil is present in small amount (1 drop) in the ginger, lavender, and orange aromatherapy inhalers. As part of the study, the participants will be asked to use an aromatherapy inhaler, which resembles a lipstick container, during three chemotherapy cycles. The participants will use the aromatherapy inhaler for 7 consecutive days. The investigators will ask the participants questions regarding demographics, clinical information, current severity of symptoms, and current methods of symptom management. There is a non-intervention baseline cycle during which subjects rate the severity of the seven different symptoms from 0 to 10 for seven consecutive days during their first chemotherapy study cycle. The next two study cycles are intervention cycles using the randomized aromatherapy. The participants will rate the severity of seven different symptoms from 0 to 10 each day the aromatherapy inhaler during one or two chemotherapy cycles (i.e., 7 consecutive days during each chemotherapy cycle). At the end of the study, the participants will be asked about his/her satisfaction with the aromatherapy used during the study. All of these measurements will provide a better understanding of the effectiveness of aromatherapy for symptom management.

DETAILED DESCRIPTION:
This study will evaluate the ability of four aromatherapy scents (ginger, lavender, orange, jojoba) to reduce the severity of seven chemotherapy-induced symptoms (nausea, vomiting, pain, anxiety/distress, fatigue, sleep difficulties, and lack of appetite). Subjects will participate in the study for two or three chemotherapy cycles. The first cycle is a non-intervention baseline cycle during which subjects rate the severity of the seven different symptoms from 0 to 10 for seven consecutive days during their first chemotherapy study cycle. The next one or two cycles are intervention cycle(s) using the assigned randomized aromatherapy. The subjects will rate the severity of seven different symptoms from 0 to 10 each day the aromatherapy inhaler during one or two chemotherapy cycles (i.e., 7 consecutive days during each chemotherapy cycle) and report if they felt the aromatherapy was helping with symptoms compared to the previous cycle. At the end of the study, the participants will be asked about his/her satisfaction with the aromatherapy used during the study. All of these measurements will provide a better understanding of the effectiveness of aromatherapy for symptom management.

ELIGIBILITY:
Inclusion Criteria:

* a) Male and female subjects, at least 8 years of age, prescribed chemotherapy for cancer. (NOTE: Only non-pregnant females are eligible). University of Rochester will enroll young adults (i.e., 21-39 years) and adults (i.e., 40 years and older). RPCI will enroll adolescents (i.e., 8-20 years) and young adults (i.e., 21-39 years).

  b) Scheduled to receive two or more cycles of chemotherapy. (NOTE: Subjects may have already started chemotherapy, but must have at least three chemotherapy cycles remaining in their current prescribed course.)

  c) Day 1 of each chemotherapy cycle must be separated from Day 1 of the next chemotherapy cycle by at least 10 days.

  d) All cancer types and chemotherapy regimens are eligible. (NOTE: Monoclonal antibody therapies are allowed if administered in combination with chemotherapy).

  e) The chemotherapy regimen must be the same regimen for all study cycles. For example, if a subject with breast cancer was prescribed TAC for Study Cycle 1, the subject must receive TAC for Study Cycles 2 and 3.

  f) Any number of chemotherapy administrations per week during a chemotherapy treatment cycle is allowed.

  g) Subjects must agree to discontinue their current use of aromatherapy for symptom management during the course of the study. They must solely use the jojoba and aromatherapy inhalers provided by the study during the course of the study.

  h) University of Rochester will enroll subjects who are able to read and understand English or Spanish. RPCI will enroll subjects who are able to read and understand English. All subjects must be able to provide informed consent in order to participate in this study.

Exclusion Criteria:

1. Subjects < 8 years old are not eligible for participation in this study.
2. Pregnant females are ineligible for the study because pregnancy is a contraindication for chemotherapy and exposure to essentials oils.
3. Subjects with more than six weeks between chemotherapy treatment cycles are not eligible.
4. Concurrent radiation therapy or interferon treatment is not allowed.
5. Subjects with any known allergy to ginger, lavender, orange, citrus of any kind, jojoba, or essential oils are not eligible.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Number of participants that complete the intervention. | 3 months
  Retention rate will be determined by arm.
Compliance rate | 3 months
  The compliance rate is the percentage of participants that report using the aromatherapy as described in protocol (i.e., at least three sniffs four times daily).

SECONDARY OUTCOMES:
Mean composite severity score | 3 months
  A composite symptom severity score will be calculated for each day during each Study Cycle. The mean composite symptom severity score will be the mean of all six composite severity scores for each cycle. We will use ANCOVA analyses to compare the maximum composite symptom severity scores and mean composite symptom severity scores between Study Cycle 3 vs Study Cycle 1 and Study Cycle 2 vs. Study Cycle 1.
Maximum composite severity score | 3 months
  The maximum composite symptom severity score will be the highest severity score across the 6 days for that cycle. The mean composite symptom severity score will be the mean of all six composite severity scores for each cycle. We will use ANCOVA analyses to compare the maximum composite symptom severity scores and mean composite symptom severity scores between Study Cycle 3 vs Study Cycle 1 and Study Cycle 2 vs. Study Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ryan Wolf, PhD, MPH, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Wilmot Canter Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
We do not currently have a plant to share individual participant data with other researchers. However, de-identified data will be shared upon request. The data shared will not contain any personal identifiers and will not be able to be linked to study subjects. Study protocol and analysis plans can be shared with other investigators upon request.